CLINICAL TRIAL: NCT02829658
Title: Use of Care Services by Patients With Borderline Personality Disorder
Acronym: EpiB
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 08 120 03
Record Dates: First submitted 2016-07-04; First posted 2016-07-12 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Psychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Psychiatric patients group: Patient groups were composed with: BPD, other PD and assessed Psychologic test
  Interventions: Behavioral: Psychologic test
- Control group: Matched controls (age, sex) composed the 3rd and 4th group (BPD control and other PD control). They were randomly chosen in the health database insurance previously used. They had no intervention.
  Interventions: Other: No intervention

INTERVENTIONS:
Behavioral: Psychologic test — Assessment by a psychologist including the Structured Interview for Diagnostic and Statistical Manual (DSM)-IV Personality Disorders (SIDP-IV) was given straight to those who had a score above 28. This questionnaire allowed us to distinguish one group of subjects with BPD and a group with other PD (without BPD). Clinical evaluation included Axis I (MINI), Axis II (SIDP-IV), psychopathological features (YSQ-I, Defense Style Questionnaire (DSQ-40), demographic variables and therapeutic alliance (Haq-II).
  Groups: Psychiatric patients group
Other: No intervention — No intervention
  Groups: Control group

SUMMARY:
Borderline personality disorder (BPD) is characterized by a pervasive pattern of instability and impulsivity. Several North American prospective studies support the high level of mental health care utilization in this population. There is little data in other systems of health organization, such as France. Furthermore, little is known on the variables associated with the mental health service utilization among BPD patients.

The main objective was to compare the utilization of mental health care among BPD patients, to the general population and patients with another personality disorder (PD) and to describe the demographic and clinical factors associated with the group of patients who use the most health care.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated with the health insurance
* Inpatient Psychiatry

Exclusion Criteria:

* Patient in forced hospitalization
* chronic psychotic disorder, mania or hypomania state, known mental retardation.
* Patient does not speak or read French

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: First, four groups were composed: BPD, other PD, control groups for PD and other PD. The first two groups were recruited from a screening of inpatients including a self-administered questionnaire (Personality Disorder Questionnaire 4+). Matched controls (age, sex) composed the 3rd and 4th group (BPD control and other PD control). They were randomly chosen in the health database insurance previously used.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2009-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Compare data among BPD Patients and general population | during five years previously to the inclusion
  Utilization of mental health care

SECONDARY OUTCOMES:
Hospitalizations | During five years previously to the inclusion
  Compare hospitalizations between BPD patients and general population
Demographics data | Inclusion
  Compare demographic data between BPD patient and general population

CONTACTS AND LOCATIONS:
Overall Officials: CAILHOL Lionel, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Cailhol L, Thalamas C, Garrido C, Birmes P, Lapeyre-Mestre M. [Mental health service utilization among borderline personality disorder patients inpatient]. Encephale. 2015 Apr;41(2):115-22. doi: 10.1016/j.encep.2014.10.008. Epub 2014 Dec 17. French. PMID 25526809